CLINICAL TRIAL: NCT06117943
Title: Pregnant Women's Knowledge of the Active and Passive Smoking Effects on Pregnancy and the Fetus
Acronym: tabac-GO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_013_tabac-GO
Record Dates: First submitted 2023-10-11; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Pregnant Women's Tabacco Exposure
Keywords: pregnancy; active smoking; passive smoking; fetus; knowledge
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women who smoke personally or are passively exposed to cigarette smoke
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — Pregnant women who smoke personally or are passively exposed to cigarette smoke

SUMMARY:
There are two remaining areas where the standards for tobacco use during pregnancy have changed little: one area is the high level of consumption by pregnant women and the other is the limited care given to pregnant women.

Indeed, many pregnant women are still over-exposed to tobacco, either through personal use or passive exposure to cigarette smoke. This passive exposure often comes from the consumption of their loved ones, such as their future co-parent or family.

However, throughout our lives, health professionals, associations, and the government send a lot of information and messages about the negative effects of tobacco on health, pregnancy, and the fetus.

This information and the possibility of receiving help from a professional trained in tobacco use exist throughout the entire pregnancy.

However, many women and their partners still do not take the necessary precautions to reduce or stop smoking. Do couples who smoke during pregnancy really have an understanding of the smoking's effects on women and their fetuses? Could they realize it and would they reduce or stop their consumption, in case they knew these negative effects?

DETAILED DESCRIPTION:
The aims are:

* To describe the knowledge of pregnant women who smoke or are exposed to tobacco smoke about the effects of active and passive smoking on the obstetrical and fetal systems.
* To identify the information that has been received by pregnant women who smoke or are confronted with tobacco smoke about the effects of tobacco on pregnancy.
* To identify information sources for pregnant women who smoke or are exposed to tobacco smoke about the negative effects of tobacco on pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women after 32 weeks of amenorrhea
* Primigravida women
* women exposed to passive or active smoking
* women aged over 18 years
* Accepting to participate in the study

Exclusion Criteria:

* Minors
* protected by law (guardianship, custodianship, judicial protection)
* refusing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women exposed to passive or active smoking.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
smoking effects on pregnancy questionnaire | day0
  Pregnant women's knowledge of the active and passive smoking effects on pregnancy : does the woman know or not risk of miscarriage, ectopic pregnancy, premature birth, premature rupture of membranes, low-lying placenta and retro-placental hematoma associated with smoking
smoking effects on the fetus questionnaire | day0
  Pregnant women's knowledge of the active and passive smoking effects on the fetus : does the woman know or not risk of premature birth, growth delay, malformation, sudden infant death syndrome associated with smoking

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Ufr Medecine Urca, Reims
  - Université de Reims Champagne Ardenne, Reims

IPD SHARING:
Plan to Share IPD: Undecided